CLINICAL TRIAL: NCT06234046
Title: Rifaximin as a Prophylaxis of Spontaneous Bacterial Peritonitis in Comparison With Ciprofloxacin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FMASU R140/2023
Record Dates: First submitted 2024-01-09; First posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Spontaneous Bacterial Peritonitis
MeSH Terms: interventions — Rifaximin; Ciprofloxacin

STUDY DESIGN:
Intervention Model Description: This randomized controlled trial was performed on two groups of Egyptian patients diagnosed with cirrhotic liver disease and ascites just recovered from SBP attack, group (1) included 40 patients were administered Rifaximin as 550 mg twice daily dosage for six months and group (2)included 40 patients were administered Ciprofloxacin as 750 mg once weekly dose for 6 months. All patients of the two groups were followed up for recurrence of SBP for 6 months.
Masking Description: no masking
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- group (1) (Active Comparator): Group (1) included 40 cases received Rifaximin as 550 mg twice daily dose for a six-months period.
  Interventions: Drug: Rifaximin 550Mg Tab; Diagnostic Test: ascitic fluid sample
- group (2) (Active Comparator): Group (2) included 40 cases received Ciprofloxacin as 750 mg once weekly dose for a six-months period.
  Interventions: Drug: Ciprofloxacin 750 MG; Diagnostic Test: ascitic fluid sample

INTERVENTIONS:
Drug: Rifaximin 550Mg Tab — group (1) received Rifaximin as 550 mg twice daily dosage for six months.
  Other Names: gastrobiotic
  Arms: group (1)
Drug: Ciprofloxacin 750 MG — group (2) received Ciprofloxacin 750 mg tab mg once weekly dosage for six months.
  Other Names: Cipro
  Arms: group (2)
Diagnostic Test: ascitic fluid sample — aspiration of ascitic fluid sample and analysis for differential cell count
  Other Names: aspiration of ascitic fluid

SUMMARY:
The goal of this Randomized controlled trial is to assessment the efficacy of Rifaximin as a prophylaxis of SBP in comparison with ciprofloxacin in Egyptian patients.

This randomized controlled trial included 80 Egyptian patients diagnosed with cirrhotic liver disease and ascites just recovered from SBP attack grouped into two groups as; Group (1) included 40 cases received Rifaximin as 550 mg twice daily dose for a six-months period and group (2) included 40 cases received Ciprofloxacin as 750 mg once weekly dose for a six-months period.

All patients of the two groups were followed up for recurrence of SBP for 6 months. The study endpoints would be SBP, death, compliance failure, or liver transplantation.

DETAILED DESCRIPTION:
This randomized controlled trial included 80 Egyptian patients diagnosed with cirrhotic liver disease and ascites just recovered from SBP attack grouped into two groups as;

* Group (1) included 40 cases received Rifaximin as 550 mg twice daily dose for a six-months period.
* Group (2) included 40 cases received Ciprofloxacin as 750 mg once weekly dose for a six-months period.

The included cases were collected from hepatology outpatient clinic and inpatient department at Ain shams University hospital between May 2023 and November 2023 after the scientific ethical committee approval. A written consent was obtained from the included cases.

Cases with metastatic HCC, patients with drug allergy from Ciprofloxacin or Rifaximin, those having ascites secondary to other causes rather than liver cirrhosis, those having gastroenterology malignancy, patients on immunotherapy, and HIV patients were all excluded from the trial. Before starting the trial, the all cases were diagnosed as SBP with ascitic fluid sample with polymorphonuclear cell count more than 250 cells /µL and received medical treatment of SBP according to EASL guidelines for treatment of SBP.

All patients of the two groups were followed up for recurrence of SBP for 6 months. The study endpoints would be SBP, death, compliance failure, or liver transplantation.

All included patients went through a comprehensive medical history, full physical assessment as well as full laboratory examination including; CBC, liver profile (ALT, AST, ALP, GGT, total & direct bilirubin, serum albumin, serum total proteins), kidney function tests (S.creat, BUN), ascitic fluid sample was taken from every patients at the starting of the trial to make sure the recovery from the previous SBP attack (AFS1) and another sample was taken once the patient was suspected to have another attack of SBP or after 6 months of treatment (AFS2). The ascitic samples were subjected to analysis of the differential cell count and measurement of ascitic albumin, glucose, total proteins and LDH, culture and sensitivity were assessed. The Child-Pugh's score were assessed, and pelvi-abdominal ultrasound were done for all patients.

ELIGIBILITY:
Inclusion Criteria:

* cirrhotic liver disease patients with ascites just recovered from SBP attack.
* Must be able to swallow tablets

Exclusion Criteria:

* Cases with metastatic HCC.
* patients with drug allergy from Ciprofloxacin or Rifaximin.
* those having ascites secondary to other causes rather than liver cirrhosis.
* those having gastroenterology malignancy.
* patients on immunotherapy.
* HIV patients.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-05-28 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
The efficacy of Rifaximin as a prophylactic treatment for SBP. | All patients of the two groups were followed up for 6 months.
  comparison between Rifaximin and Ciprofloxacin when used as a prophylaxis for the recurrence of SBP.

CONTACTS AND LOCATIONS:
Locations (1):
- Mostafa Elfors, Cairo, Egypt